CLINICAL TRIAL: NCT00001276
Title: Fasting Hypoglycemia: Diagnosis and Treatment
Brief Title: Diagnosing and Treating Low Blood Sugar Levels
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 910066; 91-DK-0066
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-11-07

CONDITIONS: Hypoglycemia; Insulinoma
Keywords: Hypoglycemia; Insulinoma; Natural History
MeSH Terms: conditions — Hypoglycemia; Insulinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hypoglycemia: Patients with hypoglycemia due to diverse etiologies.

SUMMARY:
Hypoglycemia is the term used to refer to lower than normal levels of blood sugar. This study will continue to research the causes of hypoglycemia.

Patients involved in the study will be admitted to the Clinical Center of the National Institutes of Health and undergo tests for evaluating blood sugar. Patients will be required to refrain from eating for a set period of time and will undergo blood tests for insulin levels and several other specific diagnostic tests related to insulin secretion. The patients will be under supervision and will be provided with appropriate medical and surgical attention as needed.

DETAILED DESCRIPTION:
Study Description:

The purpose of this study is to gain knowledge and experience in the diagnosis and therapy of patients with fasting hypoglycemia due to diverse etiologies, such as insulinomas. Study subjects will be evaluated and treated for their particular condition according to standard care.

Objectives:

1. To understand the pathophysiology and various causes of hypoglycemia (e.g., insulinomas, MEN1, MEN2).
2. To identify new circulating biomarkers of insulinomas.
3. To create a repository of clinical data and samples for future research of insulinomas.

Endpoints: None

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Male, females ages >= 18.
2. Patients with documented fasting blood glucose below 55 mg/dl.

4. Patients with biochemical evidence for insulinoma or other pancreatic neuroendocrine tumors.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Patients with significant cardiac disease will be excluded.
2. Subjects who are pregnant per self-report.
3. Medically unstable per the assessment of the PI.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients how are referred to us that have fasting hypoglycemia due to diverse etiologies.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 1991-05-21 (Actual)

PRIMARY OUTCOMES:
Treatment Outcomes | every 1-3 months
  resolution of hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Ranganath Muniyappa, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bar RS, Gorden P, Roth J, Siebert CW. Insulin receptors in patients with insulinomas: changes in receptor affinity and concentration. J Clin Endocrinol Metab. 1977 Jun;44(6):1210-3. doi: 10.1210/jcem-44-6-1210. PMID 194912
- [Background] Blackshear PJ, Rotner HE, Kriauciunas KA, Kahn CR. Reactive hypoglycemia and insulin autoantibodies in drug-induced lupus erythematosus. Ann Intern Med. 1983 Aug;99(2):182-4. doi: 10.7326/0003-4819-99-2-182. PMID 6349454
- [Background] Comi RJ, Gorden P. Approach to hypoglycemia in adults. Compr Ther. 1987 Mar;13(3):38-44. No abstract available. PMID 3568598
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1991-DK-0066.html